CLINICAL TRIAL: NCT02003508
Title: Prevalence of Genital HPV Infection in Males Following Introduction of Universal Male HPV Vaccination
Acronym: Impress
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marcus Chen, Adjunct Associate Professor Central Clinical School and Medical Services Manager Melbourne Sexual Health Centre, The Alfred
Other Study IDs: IISP50939
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Human Papillomavirus
Keywords: Prevalence; HPV; Human papillomavirus; Vaccination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Penile sampling for HPV DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-school based vaccination program (not vaccine eligible): Young (17-19 years) men who were not eligible for school based vaccination due to their age at the time of the programs roll out.
- Post-school based vaccination program (vaccine eligible): Young men (17-19 years) who were eligible for school based vaccination due to their age at the time of the programs roll out.

SUMMARY:
This study will examine how common HPV infection is in teenage males in Australia before and after the introduction of universal school based vaccination of males in Australia.

DETAILED DESCRIPTION:
Males aged 17 to 19 in Australia will be recruited from 2014. Men will undergo sampling from the penis for HPV. The prevalence of HPV infection will be determined in 2014-2015 and compared to the prevalence in 2016-2017.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 17 to 19
* Able to complete study requirements
* Residing in Australia from 12 years of age

Exclusion Criteria:

-Males reporting sex with males in the past 12 months

Ages: 17 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males aged 17-19 recruited from sexual health clinics and community sources
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Y Chen, PhD, Principal Investigator — Melbourne Sexual Health Centre Alfred Health and Central Clinical School Monash University
Locations (1):
- Melbourne Sexual Health Centre, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from clinical and community sources across Australia over a period of four years (February 2014- December 2017), which represented two phases. Participants recruited in phase 1 (2014-2015) were ineligible for school-based HPV vaccination. Participants in Phase 2(2016-2017) were eligible for school-based HPV vaccination.
Groups:
- Phase 1 (2014-2015): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2014-2015. This was a cohort preceding the introduction of the school-based male 4vHPV vaccination program. Accordingly, most of these men were unvaccinated against 4HPV.
- Phase 2 (2016-2017): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2016-2017. This was a cohort were age-eligible for the school-based male 4vHPV vaccination program following its introduction. Accordingly, many participants in this group had received the HPV vaccination.
Period: Overall Study
Arm/Group | Phase 1 (2014-2015) | Phase 2 (2016-2017)
Started | 179 | 166
Completed | 179 | 166
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-vaccination Period: Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2014-2015. This was a cohort preceding the introduction of the school-based male 4vHPV vaccination program.
- Post-vaccination Period: Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2016-2017. This was a cohort were age-eligible for the school-based male 4vHPV vaccination program following its introduction
- Total: Total of all reporting groups
Arm/Group | Pre-vaccination Period | Post-vaccination Period | Total
Number analyzed (Participants) | 179 | 166 | 345
Age, Continuous [Mean (Full Range); unit: years] | 18.5 [17.1 to 19.9] | 18.3 [17.1 to 19.9] | 18.4 [17.1 to 19.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 179 | 166 | 345
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 179 | 166 | 345
Sexual contact in lifetime [Count of Participants; unit: Participants] | 179 | 166 | 345

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Penile HPV Genotypes
Description: Prevalence of penile HPV genotypes among heterosexually active young men. Percentage of participants with specific genotypes on penile samples, as detected by Linear Array.
  Participants provided a single penile sample.
Time Frame: Single study visit (one time point per participant)
Population: All participants in group one were ineligible for school-based vaccination. All participants in group two were eligible to receive 4vHPV vaccination. All participants had experienced sexual contact with a female (either oral or vaginal sex), no sexual contact (either oral or anal sex) with a male, and had assessable penile samples.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 (2014-2015): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2014-2015. This was a cohort preceding the introduction of the school-based male 4vHPV vaccination program.
- Phase 2 (2016-2017): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2016-2017. This was a cohort were age-eligible for the school-based male 4vHPV vaccination program following its introduction
Arm/Group | Phase 1 (2014-2015) | Phase 2 (2016-2017)
Number analyzed (Participants) | 152 | 146
percentage of participants
  Any 4vHPV vaccine genotype | 2.6 [0.7 to 6.6] | 0.7 [0 to 3.8]
  Any of 37 HPV genotypes | 21.7 [15.4 to 29.1] | 11.6 [6.9 to 18.0]
  Any of 13 high-risk genotypes, other than 16 and 1 | 15.1 [9.8 to 21.8] | 7.5 [3.8 to 13.1]

ADVERSE EVENTS:
Time Frame: Single study visit per participant.
Groups:
- Phase 1 (2014-2015): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2014-2015. This was a cohort preceding the introduction of the school-based male 4vHPV vaccination program.
  Nil adverse events.
- Phase 2 (2016-2017): Heterosexual males aged 17-19 years, living in Australia since at least 2013. Recruited 2016-2017. This was a cohort were age-eligible for the school-based male 4vHPV vaccination program following its introduction.
  Nil adverse events.
Arm/Group | Phase 1 (2014-2015) | Phase 2 (2016-2017)
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/166
Other Adverse Events (participants affected / at risk) | 0/179 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT02003508/Prot_SAP_000.pdf